CLINICAL TRIAL: NCT04977700
Title: Using Retrospective and Real-Time Physical Activity Tracking to Predict Risk of Sunburn in Outdoor Exercisers on Strava
Brief Title: Using Physical Tracking to Predict Sunburn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0328; 1R21CA241637-01A1 (NIH)
Record Dates: First submitted 2021-07-02; First posted 2021-07-27 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Prevention
Keywords: skin cancer; physical activity
MeSH Terms: conditions — Skin Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will be enrolled on a rolling basis and participate in SS for 4 weeks in the intervention condition. After pretesting, participants will receive sun protection messages from SS through emails/comments based on results from their activity data. All participants will complete posttest survey 4 weeks from randomization.
  Interventions: Behavioral: Intervention Group
- Control Group (No Intervention): A small control group will be included to see if a no-treatment control condition is acceptable to users and estimate follow-up rates for planning a randomized trial. Participants will be enrolled on a rolling basis and will complete a pretest at randomization. All participants will complete a posttest survey 4 weeks from randomization.

INTERVENTIONS:
Behavioral: Intervention Group — Test the developed algorithm that delivers location-based, tailored sun safety advice to Strava users through Strava comments for acceptability, ways of interacting with it, and barriers/willingness to allowing access.
  Arms: Intervention Group

SUMMARY:
Recreational UV exposure is associated with every form of skin cancer and individuals who engage in more physical activity have a higher prevalence of sunburn, a proximal biomarker of melanoma risk, perhaps explaining why melanoma is the only cancer with which physical activity is positively correlated. Mobile technology for tracking physical activity has become increasingly prevalent and Strava, an activity tracking app and social networking site for athletes, is one of the most popular of these technologies. This research will test the feasibility of delivering location-based, ecologically-valid sun safety advice to Strava users at times when they are predicted to be engaged in outdoor physical activity, by utilizing Strava's public open-source Applications Programming Interface.

DETAILED DESCRIPTION:
Skin cancer is the most common cancer in the United States. Over 5.4 million cases of keratinocyte cancers (basal and squamous cell) are diagnosed annually and incidence of melanoma has increased 3% each year for the past 30 years. In the 2014 Call to Action to Prevent Skin Cancer, the U. S. Surgeon General included strategies for coordinating messages on sun safety and physical activity, recognizing the need for sun safety among populations that engage in physical activity outdoors. Recreational UV exposure is associated with every form of skin cancer; individuals who engage in more physical activity have a higher prevalence of sunburn. Melanoma is the only cancer with which physical activity is positively correlated. Strava, a tracking app and social networking site for athletes, is one of the most popular of mobile technologies for logging physical activity and providing social feedback on activities by other Strava users. The goal of this R21 research is to test the feasibility of interfacing with the Strava website and its mobile app to develop an algorithm that a) predicts when individuals are likely to be engaged in physical activity outdoors in the sun when ultraviolet radiation is high and b) delivers sun safety advice tailored to the time, location, and personal risk (e.g., skin sun sensitivity) of the Strava users. Concept focus groups with Strava users and non-users will provide input on the feasibility, content, and functions in the Strava Sun (SS) intervention. The algorithm that predicts future outdoor exercise will be developed using machine learning modeling on activity data provided by Strava users. The SS intervention will be programmed to deliver ecologically-valid sun safety advice through Strava's open-source Applications Programming Interface (API) via email and comments in the Strava interface. The sun safety advice will be tailored to location, time, season and user's personal risk, employing advice algorithms we developed for a sun safety mobile app, sunZapp, and a social media message library in our Go Sun Smart intervention for outdoor recreation resorts. SS will be tested for usability prior to conducting a pilot field trial to establish feasibility of SS in practice. The project is significant and innovative. A sun protection interface for the Strava platform will provide individuals who engage in regular physical activity personalized, ecologically-valid advice to help them practice sun safety during outdoor activities. It will contain a novel machine learning algorithm that predicts future high-risk behavior, i.e., outdoor physical activity, to provide precision prevention advice.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older; reside in the United States; read/write in English; upload outdoor activity to Strava ≥3 times per week

Exclusion Criteria:

* Younger than 18; reside outside of the United States; read/write in a language other than English; uploads Strava activity less than 3 times per week OR does not use Strava; having a cognitive or visual impairment that would interfere with participating; having another family member participating in the research; having participated in the focus group and usability testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Berteletti, MSW, Principal Investigator — Klein Buendel, Inc.
Locations (1):
- Klein Buendel, Inc., Golden, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: n=123 participants were recruited and screened for participation in formative research prior to the pilot study detailed, including focus groups, usability testing, and collection of activity data. None of those participants were randomized. n=41 participants participated in the randomized pilot as described in this entry.
Groups:
- Intervention Group: Participants will be enrolled on a rolling basis and participate in SS for 4 months in the intervention condition. After pretesting, participants will receive sun protection messages from SS through emails/comments based on algorithm results from their profile and activity data. All participants will complete posttest survey 4 months from randomization.
  Intervention Group: Test the developed algorithm that delivers location-based, tailored sun safety advice to Strava users through Strava comments for acceptability, ways of interacting with it, and barriers/willingness to allowing access.
- Control Group: A small control group will be included to see if a no-treatment control condition is acceptable to users and estimate follow-up rates for planning a randomized trial. Participants will be enrolled on a rolling basis and will complete a pretest at randomization. All participants will complete a posttest survey 4 months from randomization.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 31 | 10
Completed | 31 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants are adults in the United States who exercise outdoor and use the Strava platform to log activity data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 31 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 7 | 35
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (14.8) | 48.9 (17.9) | 43.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 7 | 29
  Male | 9 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 31 | 9 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 26 | 10 | 36
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Sun Protection Practices
Description: What proportion of 8 sun protection practices did participants do on reported days of exercise. Participants responded to 8 potential sun protection practices and provided the number of days they did each practice within the timeframe provided (3 months at baseline; 4 weeks at posttest). Participants also provided number of days of outdoor exercises within timeframe. Proportion was calculated by dividing the frequency of each sun protection practice by the number of days of outdoor exercise within the timeframe. Mean score of all sun protection practices per day of outdoor exercise is reported. Range = 0-1, where a higher number indicates more sun safety practices performed. A proportion was used to account for different timeframes at baseline and posttest.
Time Frame: baseline and four-weeks post intervention
Measure: Mean (Standard Deviation); unit: proportion of practices/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
proportion of practices/day
  baseline | 0.30 (0.35) | 0.43 (0.43)
  four week posttest | 0.35 (0.37) | 0.41 (0.45)

2. Primary Outcome: Prevalence of Sunburn
Description: Participants were asked if their skin was sunburned (described as being red and/or painful from exposure to the sun) in the past three months, and if so, how many times.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: sunburn
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
sunburn | 1.0 (2.7) | 0.2 (0.6)

3. Primary Outcome: Prevalence of Sunburn
Description: Participants were asked if their skin was sunburned (described as being red and/or painful from exposure to the sun) in the past four weeks, and if so, how many times.
Time Frame: four-weeks post intervention
Measure: Mean (Standard Deviation); unit: sunburn
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
sunburn | 0.3 (0.6) | 0.3 (0.7)

4. Secondary Outcome: Physical Activity (Godin Leisure-Time Exercise Questionnaire)
Description: Duration in minutes of exercise multiplied by number of times per week, in the past 7 days. Total minutes per week calculated; mean per treatment group reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
minutes | 578.1 (603.3) | 465.8 (250.4)

5. Secondary Outcome: Physical Activity (Godin Leisure-Time Exercise Questionnaire)
Description: as for outcome 4
Time Frame: four-weeks post intervention
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
minutes | 474.6 (238.4) | 657.5 (578.0)

6. Secondary Outcome: Recall of Sun Protection Messages
Description: Participants in intervention only were asked about how many messages they read. Scale ranges from 0 - 3. 0 = none of the messages; 1 = some of the messages; 2 = most of the messages; 3 = all of the messages. Higher score indicates higher message recall.
Time Frame: four weeks post intervention
Population: Control group participants were not given this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 0
units on a scale | 1.9 (1.0) |

7. Secondary Outcome: Self-Efficacy for Sun Protection When Exercising
Description: Participants were asked: how confident are you that you can practice sun safety next time that you exercise. 1 = not confident; 2 = a little confident; 3 = somewhat confident; 4 = very confident. Higher scores indicates more self-efficacy for sun safety.
Time Frame: baseline and four-weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
units on a scale
  baseline | 3.1 (0.9) | 3.4 (0.8)
  four-week follow-up | 3.4 (0.8) | 3.3 (0.5)

8. Secondary Outcome: Range of Physical Activity (Godin Leisure-Time Exercise Questionnaire)
Description: as for outcome 4
Time Frame: baseline
Measure: Mean (Full Range); unit: minutes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
minutes | 578.1 [36 to 2580] | 465.8 [138 to 960]

9. Secondary Outcome: Range of Physical Activity (Godin Leisure-Time Exercise Questionnaire)
Description: as for outcome 4
Time Frame: four weeks post-intervention
Measure: Mean (Full Range); unit: minutes
Groups:
- Intervention Group: Participants will be enrolled on a rolling basis and participate in SS for 4 weeks in the intervention condition. After pretesting, participants will receive sun protection messages from SS through emails/comments based on algorithm results from their profile and activity data. All participants will complete posttest survey 4 weeks from randomization.
  Intervention Group: Test the developed algorithm that delivers location-based, tailored sun safety advice to Strava users through Strava comments for acceptability, ways of interacting with it, and barriers/willingness to allowing access.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 10
minutes | 474.6 [0 to 1020] | 657.5 [285 to 2220]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/10
Other Adverse Events (participants affected / at risk) | 0/31 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04977700/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04977700/ICF_001.pdf